CLINICAL TRIAL: NCT03573843
Title: Cognitive Stimulation Guided by a Software to Prevent Delirium in Older Patients
Brief Title: Software-guided Cognitive Stimulation to Prevents Delirium
Acronym: Prevedel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Tobar, Associated professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCHID16AM0080
Record Dates: First submitted 2018-05-04; First posted 2018-06-29 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Delirium in Old Age
Keywords: Delirium; Prevention; Cognitive stimulation
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Patients who meet the inclusion / exclusion criteria will be randomly assigned to the Control group: They will continue to receive the standard prevention measures: delirium detection, treatment health team education and the patient's family, sleep hygiene plan, early mobilization , resolve sensorial deterioration, and delivery of information of temporal-spatial reorientation in a continuous manner, plus the use of a mobile device without installed delirium prevention software (placebo).
  Interventions: Other: Placebo
- Experimental (Experimental): Patients who meet the inclusion / exclusion criteria will be randomly assigned to the experimental group:They will continue to receive standard prevention measures: Detection of delirium, education of health care team and the patient's family, sleep hygiene plan, early mobilization, resolve sensory impairments, and delivery of information of temporal-spatial reorientation in continuously, plus the use of software installed on a mobile device designed to support the prevention of delirium (Prevention software).
  Interventions: Other: Prevention software

INTERVENTIONS:
Other: Prevention software — All patients will have a tablet with the software PREVEDEL between 09:00-19:00 hrs.
  Arms: Experimental
Other: Placebo — All patients will have a tablet without the software PREVEDEL between 09:00-19:00 hrs.
  Arms: Control

SUMMARY:
This study is a pilot randomized controlled trial, comparing a group of older patients with standardized non-pharmacological delirium prevention plus a basic tablet versus a group with standardized non-pharmacological delirium prevention plus a tablet with a software of cognitive stimulation (PREVEDEL).

Software:It is a local development, including a interprofessional team of delirium healthcare experts, older patients and a team og engineers. The software was developed during the first year of this project and was inscribed for author rights.

Inclusion criteria: Older patients > 65 y.o. Admitted to medicine room or intermediate care unit > 48 hrs, and informed consent to participate.

Exclusion Criteria:Delirium positive, neuroleptic use, dementia, and non-spanish speakers.

The study was approved by ethical committee of Hospital Clinico University of Chile Standardized Non-pharmacological intervention: Health workers were previously educated in delirium, and environmental issues were implemented. This intervention coverage in nine different domains: orientation, early mobilization, environmental noise and light, sensorial deficit, sleep, hydratation, drug reduction, and family participation.

Intervention: All patients will have a tablet with or without the software PREVEDEL between 09:00-19:00 hrs.

Measures: delirium will be monitoring with CAM (Confusion Assessment Method) twice a day for 5 days.

Primary outcome: Delirium rate between both groups Secondary outcomes:Long of stay, severity od delirium, time of use of electronic device, and Barthel to discharge.

ELIGIBILITY:
Inclusion Criteria:

Older patients > 65 y.o. Admitted to medicine room or intermediate care unit > 48 hrs, and informed consent to participate.

Exclusion Criteria:

Delirium positive, neuroleptic use, dementia, and non-spanish speakers.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Difference in delirium incidence between both groups | 5 days
  Delirium will be assessed with CAM (the confusion assessment method) twice a day.

SECONDARY OUTCOMES:
Length of stay | 5 days
  The days of total hospital stay of the patients will be recorded
Severity of delirium | 5 days
  Delirium will be evaluated with CAM-S (the confusion assessment method Severity) whenever appropriate.
Time of use of electronic device | 5 days
  The usage time on the mobile device (with internal device registration) will be recorded.
Functionality at discharge. | 5 days
  Functionality at discharge will be assessed with Barthel Index test at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo A Tobar, MD, Study Director — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, International, Chile

IPD SHARING:
Plan to Share IPD: No